CLINICAL TRIAL: NCT05570539
Title: A Phase 1, Single-Centre, Open-Label, Two-Part, Sequential Cross-Over Study Designed to Assess the Pharmacokinetic Profile of BLU-5937 Following Administration of Extended Release Formulation Prototypes and an Immediate Release Reference Formulation in Healthy Male and Female Subjects
Brief Title: Assessment of the Pharmacokinetics of BLU-5937 Extended Release Prototypes and a BLU-5937 Immediate Release Reference Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 222418; BUS-P1-09 (Other: Bellus Health Inc)
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cough; Healthy
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate Release formulation (Active Comparator): IR Formulation
  Interventions: Drug: BLU-5937 IR
- Extended Release formulation (Experimental): ER formulation
  Interventions: Drug: BLU-5937 ER

INTERVENTIONS:
Drug: BLU-5937 IR — Each subject will receive two single and multiple administrations of Immediate Release reference formulation
  Arms: Immediate Release formulation
Drug: BLU-5937 ER — Each subject will receive single and multiple oral administrations of Extended Release formulation
  Arms: Extended Release formulation

SUMMARY:
This is a Phase 1, Single-Centre, Open-Label, Two-Part, Sequential Cross-Over Study Designed to Assess the Pharmacokinetic Profile of BLU-5937 Following Administration of Extended Release Formulation Prototypes and an Immediate Release Reference Formulation in Healthy Male and Female Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females

Exclusion Criteria:

* History of clinically significant cardiovascular, renal, hepatic, metabolic, dermatological, respiratory, GI, neurological, endocrine, haematological, immunological or psychiatric disorder, as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Measurement of the maximum observed plasma drug concentration (Cmax) | Pre dose up to 36 hours post-dose
  To assess the comparison between Cmax following administration of an Extended Release tablet formulation and an Immediate Release reference formulation.
Measurement of the minimum observed plasma drug concentration (Cmin) | Pre dose up to 36 hours post-dose
  To assess the comparison between Cmin following administration of an Extended Release tablet formulation and an Immediate Release reference formulation.
Measurement of the area under the plasma drug concentration by time curve AUC | Pre dose up to 36 hours post-dose
  To assess the comparison between AUC following administration of an Extended Release tablet formulation and an Immediate Release reference formulation.
Measurement of the observed plasma drug concentration 24 hours post-dose (C24) | 24 hours post-dose
  To assess the comparison between C24 following administration of an Extended Release tablet formulation and an Immediate Release reference formulation.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No